CLINICAL TRIAL: NCT03472898
Title: The Unidentified Association of Gated SPECT Abnormality With J Point Elevation
Brief Title: Gated SPECT Abnormality With J Point Elevation
Status: Completed | Type: Observational
Sponsor: Ankara Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Aylin AKBULUT, University of Health Sciences Ankara Training and Research Hospital, Ankara Education and Research Hospital
Other Study IDs: 0001
Record Dates: First submitted 2018-03-15; First posted 2018-03-21 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Cardiovascular Diseases; Electrocardiogram: Electrical Alternans; Myocardial Ischemia; Early Repolarization Syndrome; Left Ventricular Hypokinesia
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators present an interesting co-incidence of Gated wall abnormality in the inferolateral wall in normal sestamibi myocardial perfusion images with J wave in the inferior derivations of the ECG in a patient. The subsequent coronary angiography demonstrated 80% mid right coronary artery (RCA) stenosis, which was intervened with a drug-eluting stent. The investigators conclude that even though the myocardial perfusion is normal, the association of gated wall abnormality with J wave presentation within the same location should be further evaluated.

DETAILED DESCRIPTION:
The isolated J-point elevation considered as a type of "early repolarization" pattern (ER), is commonly been regarded as a benign finding. However, ER associations with arrhythmic sudden death from CAD or sudden cardiac death due to either idiopathic ventricular fibrillation have been shown. A recent study reported that ER especially in inferior leads, was related to worse cardiac outcomes in patients with CAD and they argue that ER in patients with CAD seems to be associated with the myocardial scar in the absence of pathologic Q waves.

Likewise, it is rare to detect clinically important gated SPECT abnormalities in normal myocardial perfusion studies with normal transient ischemic dilatation (TID) score and without any right ventricular uptake or any pulmonary uptake. Normal myocardial perfusion findings with wall motion abnormalities are frequently encountered in the interventricular septum of the patients who have previous bypass surgery or in patients with left bundle branch block (LBBB). However, the presented patient did not have the history of any intervention or LBBB. Perfusion and function discordance can be encountered in non-ischemic dilated cardiomyopathy patients; nonetheless, EF is markedly reduced in these patients.

The presented case, J point elevation in the ECG associated with relative wall motion abnormality was an important clue to determine CAD in the lack of evident perfusion defects or significant ECG findings.

The presence of wall motion abnormalities during stress study to predict CAD in patients with normal perfusion pattern, owing to balanced ischemia, was not only reported in multi-vessel disease but also in single-vessel disease without having presented the association between either regional wall motion abnormality or a localized particular ECG pattern and culprit lesion territory.

The interesting part of the presented case is, notwithstanding the myocardial perfusion pattern is normal, the abnormal gated finding with ECG changes having the concordant localization can be a significant milestone on the way to the diagnosis. To the best of investigators knowledge, the association between J point elevation and wall motion abnormality have not been described yet. Therefore, the investigators would like to draw attention to the importance of adjoining trivial ECG changes and wall motion abnormality for readers anymore.

ELIGIBILITY:
Inclusion Criteria:

* Case Report

Exclusion Criteria:

* None

Ages: 55 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Case Report
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2018-01-17 (Actual); Study Completion 2018-01-17 (Actual)

PRIMARY OUTCOMES:
Case Report Proposal | December 2017-January 2018
  Cure

CONTACTS AND LOCATIONS:
Overall Officials: Aylin Akbulut, Study Chair — Ankara Education and Research Hospital
Locations (1):
- AnkaraERH, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No